CLINICAL TRIAL: NCT03344965
Title: A Phase 2 Study of Olaparib Monotherapy in Metastatic Breast Cancer Patients With Germline or Somatic Mutations in DNA Repair Genes (Olaparib Expanded)
Brief Title: Olaparib In Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Johns Hopkins University (Other); AstraZeneca (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nadine Tung, Prinicipal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-428
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer; Invasive Breast Cancer; Somatic Mutation Breast Cancer (BRCA1); Somatic Mutation Breast Cancer (BRCA2); CHEK2 Gene Mutation; ATM Gene Mutation; PALB2 Gene Mutation; RAD51 Gene Mutation; BRIP1 Gene Mutation; NBN Gene Mutation
Keywords: Metastatic Breast Cancer; Invasive Breast Cancer; Somatic Mutation Breast Cancer (BRCA1); Somatic Mutation Breast Cancer (BRCA2)
MeSH Terms: conditions — Breast Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- OLAPARIB QD GERMLINE MUTATION (Experimental): After the screening procedures confirm eligibility to participate in the research study:
  * Olaparib: Each study treatment cycle lasts 21 days (3 weeks), taking 2 times per day, 12 hours apart.
  * Tumor measurement q6 weeks x 24 weeks, then q 12 weeks
  Interventions: Drug: Olaparib
- OLAPARIB QD GERMLINE MUTATION - EXPANSION (Experimental): After the screening procedures confirm eligibility to participate in the research study:
  * Olaparib: Each study treatment cycle lasts 21 days (3 weeks), taking 2 times per day, 12 hours apart.
  * Tumor measurement q6 weeks x 24 weeks, then q 12 weeks
  Interventions: Drug: Olaparib
- OLAPARIB QD SOMATIC MUTATION (Experimental): After the screening procedures confirm eligibility to participate in the research study:
  * Olaparib: Each study treatment cycle lasts 21 days (3 weeks), taking 2 times per day, 12 hours apart.
  * Tumor measurements q6 weeks x 24 weeks, then q 12 weeks
  Interventions: Drug: Olaparib
- OLAPARIB QD SOMATIC MUTATION - EXPANSION (Experimental): After the screening procedures confirm eligibility to participate in the research study:
  * Olaparib: Each study treatment cycle lasts 21 days (3 weeks), taking 2 times per day, 12 hours apart.
  * Tumor measurements q6 weeks x 24 weeks, then q 12 weeks
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — olaparib tablets bid daily continuously on a 21 day cycle until progression, intolerable toxicity, consent withdrawn, patient noncompliance or death.
  Other Names: AZD2281; KU-0059436

SUMMARY:
This research study is for patients with metastatic breast cancer.

* Metastatic means that the cancer has spread beyond the breast. In addition, through genetic testing of the blood or tumor, an altered gene has been found that suggests the tumor may not be able to repair its genetic material (DNA) when it becomes damaged.
* This aspect of the cancer may cause it to be more sensitive - that is, more effectively killed by certain types of drugs such as the study agent being evaluated in this trial, Olaparib.

  * Olaparib is a type of drug known as a PARP inhibitor. Some types of breast cancer and ovarian cancer share some basic features that make them sensitive to similar treatments. Information from those other research studies suggests that this drug may help to treat metastatic breast cancer.

    * This study will evaluate whether olaparib is effective in breast cancer patients whose tumor has a mutation in one of the other genes that function with BRCA1 and BRCA2 to repair damaged DNA .This mutation may have been inherited from a parent, or may have developed only in the tumor.
    * This study will also evaluate whether olaparib is effective in breast cancer patients whose tumor has a mutation in BRCA1 or BRCA2 that was acquired by the tumor, but not inherited.

DETAILED DESCRIPTION:
* This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the study drug, Olaparib, is being studied for use in this setting and the research doctors are trying to learn more about it-the side effects it may cause and if the drug is effective in treating this type of cancer.
* What is a DNA repair gene mutation?

  -- In order to survive, all cells, even cancer cells, must be able to repair their genetic material (DNA) when it gets damaged. A mutation is an alteration or change in a gene- either inherited from a parent or acquired over time- that prevents the gene from working properly. Faulty genes (or genes that carry a mutation) have been linked to increased risk of hereditary breast and ovarian cancer.
* What is Olaparib?

  * Olaparib is a drug that may stop cancer cells from growing. Olaparib is a PARP inhibitor which means that it blocks an enzyme (proteins that help chemical reactions in the body occur) in cells called PARP. PARP helps repair DNA when it becomes damaged. It has been shown that the tumors in individuals who have inherited or acquired a mutation in the BRCA1 or BRCA2 genes are often sensitive to killing by PARP inhibitors.
  * In normal cells and many other tumors, repair of damage to the DNA requires pathways of genes that work with BRCA1 and BRCA2. Therefore, when a drug that inhibits PARP from working is given to people with a BRCA mutation, or a defect in another gene that works with BRCA1 and BRCA2, both ways of repairing damaged DNA no longer work. The combined effect of knocking out both DNA repair mechanisms is so severe that the cancer cells could die. This might stop the growth of type of breast cancer, but this is not known.
  * The FDA (U.S. Food and Drug Administration) has approved Olaparib for use in advanced ovarian cancer with a BRCA1 or BRCA2 mutation. Olaparib is not approved for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed invasive breast cancer with stage IV disease, either biopsy proven or with unequivocal evidence of metastatic disease by physical examination or radiological study.
* Cohorts 1 and 2: Documented germline (Cohort 1) or somatic mutation or homozygous deletion (Cohort 2) in one of the DNA repair genes listed below that is deleterious or suspected to be deleterious, and no germline BRCA1 or BRCA2 mutation. The mutation may be identified through any CLIA approved NGS panel.

  * ATM, ATR, BARD1, BRIP1 (FANCJ), CHEK2 , FANCA, FANCC, FANCD2, FANCE, FANCF, FANCM, MRE11A, NBN, PALB2, RAD50, RAD51C, RAD51D, plus other HR-related genes at the discretion of Dr. Tung with the key study collaborators (see details below in italics). (Cohorts 1 or 2)

    --- OR
  * Documented somatic mutation (deleterious or suspected deleterious) in BRCA1 or BRCA2 through any CLIA approved lab only if in addition to the lack of a germline BRCA1/2 mutation is demonstrated through a CLIA approved lab. Patients with germline mutations in BRCA1/2 are NOT eligible for this study. (Cohort 2 only)
* Cohort 1a: germline PALB2 mutation

  -- The mutation must be identified through a CLIA-approved NGS panel. Mutations must be reviewed and confirmed by Dr. Tung to meet eligibility prior to registration.
* Cohort 2a: somatic mutation of BRCA 1 or BRCA 2

  -- The mutation must be identified through a CLIA-approved NGS panel. Mutations must be reviewed and confirmed by Dr. Tung to meet eligibility prior to registration. Documentation of absence of germline mutation in BRCA 1/2 is required.
* All deep (homozygous) deletions, frameshift mutations and truncating mutations in the genes listed above are eligible as well as missense variants in these genes that have previously been reported as pathogenic or likely pathogenic. If there is a discrepancy between two labs regarding the pathogenicity of a particular variant, the final decision regarding eligibility will be determined by the study steering committee.
* At least one measurable lesion that can be accurately assessed at baseline by CT (MRI where CT is contraindicated) and is suitable for repeated assessment as per RECIST 1.1.

  -- NOTE: If the only site of measurable of disease has been previously irradiated, there must be evidence of post-radiation progression. For a lesion to be considered as measurable, it must be one that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements
* Patients may not have progressed on more than two chemotherapy regimens in the metastatic setting.
* The following will NOT be counted as a prior line of cytotoxic chemotherapy:

  * If a patient discontinued a cytotoxic regimen due to toxicity (e.g., hypersensitivity or neuropathy) but had not progressed on that regimen, or if a prior chemotherapy regimen was discontinued after response achieved, it will not be counted in the number of prior chemotherapy regimens allowed.
  * Prior hormonal therapy and non-hormonal targeted therapy; including the combination of an aromatase inhibitor and everolimus.
  * Targeted and biologic therapies.
  * The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as this was started at least 5 days prior to study treatment.
* The most recent cytotoxic, biologic or targeted therapy received must have been completed at least 21 days prior to study treatment; hormonal therapy must have been completed at least 7 days prior, unless otherwise noted.
* Prior therapy is allowed as follows:

  * Platinum chemotherapy in the adjuvant setting is allowed, if the last platinum dose was > 12 months before identification of metastatic disease. Platinum-based chemotherapy in the metastatic setting is not permitted.
  * History of prior anthracycline (e.g. doxorubicin, epirubicin) and taxane-based (e.g. paclitaxel, docetaxel) chemotherapy in the neo-adjuvant / adjuvant or metastatic setting is preferred, but not required.
  * Patients with hormone receptor-positive (estrogen and/or progesterone receptor-positive) disease must have received and progressed on at least one endocrine therapy (adjuvant or metastatic), or have disease that the treating physician believes to be inappropriate for endocrine therapy. Endocrine therapy must have been completed at least 7 days before study treatment.
  * Prior radiation is allowed; radiation therapy must have been completed at least 21 days before study treatment.
  * Prior treatment with FDA approved or investigational biologics (other than PARP inhibitors) and novel molecularly targeted therapies, including oral or IV formulations, shall not exclude patients from participation.
  * For agents with ambiguous categorization, final determination of patient eligibility will be made by the Protocol Chair prior to enrollment.
  * Prior PARP inhibitor use is not allowed for this study
* Age ≥ 18 years.
* ECOG performance status 0-1 (Karnofsky ≥60%, see Appendix A) Life expectancy ≥16 weeks
* Participants must have normal organ and bone marrow function measured within 28 days prior to registration as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * white blood cells > 3,000/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥ 10.0 g/dL with no blood transfusions (packed red blood cells in the past 28 days is permitted)
  * total bilirubin ≤ 1.5 x institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Serum or plasma creatinine ≤ 1.5 x institutional upper limit of normal (ULN)

    --- OR
  * creatinine clearance ≥51 mL/min/1.73 m2 for participants
  * Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72 ---- a where F=0.85 for females and F=1 for males.
* Willingness to undergo biopsy.
* Patients with a history of treated CNS metastases are eligible, provided they meet all of the following criteria: Disease outside the CNS is present; no clinical evidence of progression since completion of CNS-directed therapy; minimum of 2 weeks between completion of radiotherapy and Cycle 1 Day 1 and recovery from significant (Grade ≥3) acute toxicity with no ongoing requirement for > 10mg of prednisone per day or an equivalent dose of other corticosteroid. NOTE: Patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
* Both men and women are eligible for this study
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential. For women who are not post-menopausal, a negative urine or serum pregnancy test is required within 28 days of study treatment and confirmed prior to treatment on day 1.
* Post-menopausal is defined as one of the following:

  * > 60 years old
  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
  * radiation-induced oophorectomy with last menses >1 year ago
  * surgical sterilisation (bilateral oophorectomy or hysterectomy)
* Men and women of reproductive potential need to employ two highly effective and acceptable forms of contraception throughout their participation in the study and for 30 days (for women) or 90 days (for men) after the last dose of study medication because the effects of olaparib on the developing human fetus are unknown. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Ability to understand and the willingness to sign a written informed consent document. Informed consent must be provided prior to any study specific procedures

Exclusion Criteria:

* Any previous treatment with a PARP inhibitor, including olaparib.
* Germline BRCA1 or BRCA2 mutation
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) and grapefruit, grapefruit juice or any product containing grapefruit,or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Persistent toxicities (≥CTCAE grade 2) caused by previous cancer therapy, excluding alopecia
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with prior myelodysplastic syndrome or acute myeloid leukemia.
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer; curatively treated in situ cancer of the cervix; ductal carcinoma in situ (DCIS); Stage 1, grade 1 endometrial carcinoma; or, other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years
* Resting EKG with QTc > 470 msec or family history of long QT syndrome. If EKG demonstrates QTc >470 msec, patient will be eligible only if repeat EKG demonstrates QTc ≤470 msec.
* Pregnant or breast feeding women.
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Major surgery within 2 weeks of starting study treatment: patients must have recovered from any effects of any major surgery.
* Patients with known active hepatitis (i.e., Hepatitis B or C)
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 21 Days
  RECIST 1.1 criteria will be reported with a two-sided 90% confidence interval using the method from Atkinson and Brown to account for the two-stage design

SECONDARY OUTCOMES:
Clinical Benefit Rate | 16 weeks
  Reported with 90% binomial exact confidence intervals.
Progression Free Survival | 36 Months
  Kaplan-Meier
Stable Disease | 36 Months
  Kaplan-Meier
Number of Participants with Severe Adverse Events | after the first dose of study treatment and ends 30 days following the last administration of study treatment or study discontinuation/termination,
  Treatment-related toxicities will be summarized within and across Cohorts by maximum grade and by term using CTCAE v4.0 and reported with 90% binomial exact confidence intervals.
Mutant Allele Frequency | 36 months
  Two-sample t-test with 10% Type-I error level

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Tung, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center Westchester, East White Plains, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center Nassau, Uniondale, New York
  - Duke University, Durham, North Carolina
  - UPMC Hillman Cancer Center - Erie, Erie, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington Fred Hutchinson Cancer Care, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tung NM, Robson ME, Ventz S, Santa-Maria CA, Nanda R, Marcom PK, Shah PD, Ballinger TJ, Yang ES, Vinayak S, Melisko M, Brufsky A, DeMeo M, Jenkins C, Domchek S, D'Andrea A, Lin NU, Hughes ME, Carey LA, Wagle N, Wulf GM, Krop IE, Wolff AC, Winer EP, Garber JE. TBCRC 048: Phase II Study of Olaparib for Metastatic Breast Cancer and Mutations in Homologous Recombination-Related Genes. J Clin Oncol. 2020 Dec 20;38(36):4274-4282. doi: 10.1200/JCO.20.02151. Epub 2020 Oct 29. PMID 33119476